CLINICAL TRIAL: NCT03428178
Title: Efficacy Study of Gene Therapy for The Treatment of Acute LHON Onset Within Three Months
Acronym: LHON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bin Li (Other)
Responsible Party: Sponsor-Investigator, Bin Li, Clinical Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LHON(Acute)
Record Dates: First submitted 2018-01-07; First posted 2018-02-09 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Acute LHON; Onset Within Three Months; Onset Between 3 to 6 Months; Onset Between 6 to 12 Months; Onset Between 12 to 24 Months; Onset Between 24 to 60 Months; Onset Over 60 Months
Keywords: Acute LHON; onset within three months; onset between 3 to 6 months; onset between 6 to 12 months; onset between 12 to 24 months; onset between 24 to 60 months; onset over 60 months

STUDY DESIGN:
Intervention Model Description: 20 patients of Leber Hereditary Optic Neuropathy (LHON) onset within 3 months,20 between 3 to 6 months,20 between 6 to 12 months,20 between 12 to 24 months,20 between 24 to 60 months,and 20 over 24 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rAAV2-ND4 (Experimental): A Single IVT of recombinant Adeno-Associated Virus-NADH dehydrogenase, subunit 4 (complex I)（rAAV2-ND4)（0.05ml).The dose is 1 × 10^10 vg/0.05 mL for test groups.
  Interventions: Drug: rAAV2-ND4

INTERVENTIONS:
Drug: rAAV2-ND4 — rAAV2-ND4 of vitreous cavity injection
  Other Names: rAAV2-ND4 gene therapy

SUMMARY:
Efficacy Study of Gene Therapy for The Treatment of Acute Leber's Hereditary Optic Neuropathy (LHON) onset within three months

DETAILED DESCRIPTION:
Leber's Hereditary Optic Neuropathy (LHON) is a maternally inherited ocular disorder associated with a mutation in mtDNA .The disease is a common cause of teenaged blindness in both eyes for which there is currently no effective treatment.

In 2008, the investigators recognized that gene therapy for LHON could be performed not only theoretically but technically. The investigators have been carring out a series of basic and clinical studies from constructing the vectors to identifying and mitigating safety issues . After performing several animal experiments, the investigators had moved into clinical trials. In 2011, the investigators performed the first LHON gene therapy trial in the world, which was registered in December 2010 at ClinicalTrials.gov (Registration number: CT01267422) and was a preliminary study to verify the safety and efficacy of gene therapy for LHON . In the 36-month follow-up, the investigators found that six out of nine patients have vision improvement obviously and no adverse events were observed.

This is a multi - center , prospective study of 120 patients with the G11778A mutation in Mt-DNA.This clinical trial recruited 20 patients with the 11778 mutation of MT-DNA onset within three months,20 between 3 to 6 months,20 between 6 to 12 months,20 between 12 to 24 months,20 between 24 to 60 months,and 20 over 60 months.. All patients will be treated with a Single vitreous cavity injection of recombinant Adeno-Associated Virus-NADH dehydrogenase, subunit 4 (complex I)（rAAV2-ND4)（0.05ml), with dose 1 × 10^10 vg/0.05 mL .The eye of treatment is up to the time of onset.

The visual acuity, visual field,visual evoked potential （VEP）,optical coherence tomography（ OCT）, electroretinograms(ERG), retinal nerve fiber layer(RNFL)and Liver and kidney function in plasma were compared after treatment at 1,2,3,6and 12 months interval.

ELIGIBILITY:
Inclusion Criteria:

1. Patients carry the mitochondrial point mutation at 11778, which is consistent with the diagnostic criteria for LHON.
2. The vision falls within 3 months,onset between 3 to 6 months,onset between 6 to 12 months,onset between 12 to 24 months,onset between 24 to 60 months,and onset over 60 months.
3. Patients signed written informed consent.
4. Patients are between the ages of 8 and 60 years old and able to tolerate the gene therapy procedure which includes local anesthesia.
5. Patients are willing to follow the doctor's instructions and to consult the doctor at prescribed times.
6. Patient's physical examination results are all normal, including liver function, kidney function, routine blood test, routine urine test, complete immunological test, and humoral immune response.

Exclusion Criteria:

1. Patients who are wearing a cardiac pacemaker, suffering from severe heart, lung or kidney function failure, various hemorrhagic diseases, acute infectious diseases, high fever, or convalescing after heart surgery or who are pregnant are excluded.
2. Patients who are participating in other clinical studies are excluded.
3. Patients who suffer from a diagnosed mental problem are excluded.
4. Patients who suffer from chronic diseases such as diabetes and hypertension are excluded.
5. Patients who show abnormal test results such as positive AAV2 humoral immune response (positive means that the AAV2 neutralizing antibody assay of patient was significant different when comparing free serum with 1:20 serum concentrations) and abnormal human T lymphocyte subsets CD3+, CD3+/CD4+ and CD3+/CD8+ prior to gene therapy surgery are excluded.

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
BCVA | Change from Baseline at 12 months
  The Best Corrected Visual Acuity

SECONDARY OUTCOMES:
Computerized Visual Field | Change from Baseline at 12 months
  Visual Field index
Computerized Visual Field | Change from Baseline at 12 months
  Mean Defect
VEP | Change from Baseline at 12 months
  visual evoked potential
RNFL | Change from Baseline at 12 months
  retinal nerve fiber layer
Liver function in plasma | Before treatment and in the first ,third,sixth,twelfth month after the treatment
  Before and after the treatment,Liver function in plasma will be checked.
kidney function in plasma | Before treatment and in the first ,third,sixth,twelfth month after the treatment
  Before and after the treatment,kidney function in plasma will be checked.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology ，Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang S, Ma SQ, Wan X, He H, Pei H, Zhao MJ, Chen C, Wang DW, Dong XY, Yuan JJ, Li B. Long-term outcomes of gene therapy for the treatment of Leber's hereditary optic neuropathy. EBioMedicine. 2016 Aug;10:258-68. doi: 10.1016/j.ebiom.2016.07.002. Epub 2016 Jul 6. PMID 27426279
- [Background] Yang S, Yang H, Ma SQ, Wang SS, He H, Zhao MJ, Li B. Evaluation of Leber's hereditary optic neuropathy patients prior to a gene therapy clinical trial. Medicine (Baltimore). 2016 Oct;95(40):e5110. doi: 10.1097/MD.0000000000005110. PMID 27749593
- [Background] Ran R, Yang S, He H, Ma S, Chen Z, Li B. A retrospective analysis of characteristics of visual field damage in patients with Leber's hereditary optic neuropathy. Springerplus. 2016 Jun 23;5(1):843. doi: 10.1186/s40064-016-2540-7. eCollection 2016. PMID 27386292
- [Background] Wan X, Pei H, Zhao MJ, Yang S, Hu WK, He H, Ma SQ, Zhang G, Dong XY, Chen C, Wang DW, Li B. Efficacy and Safety of rAAV2-ND4 Treatment for Leber's Hereditary Optic Neuropathy. Sci Rep. 2016 Feb 19;6:21587. doi: 10.1038/srep21587. PMID 26892229
- [Background] Yang S, He H, Zhu Y, Wan X, Zhou LF, Wang J, Wang WF, Liu L, Li B. Chemical and material communication between the optic nerves in rats. Clin Exp Ophthalmol. 2015 Nov;43(8):742-8. doi: 10.1111/ceo.12547. Epub 2015 Jun 25. PMID 25950380
- [Background] Pei H, Wan X, Hu W, Dong X, Li B. Construction and detection of a novel type of recombinant human rAAV2/2-ND4. Eye Sci. 2013 Jun;28(2):55-9. PMID 24396955
- [Background] Cui G, Ding H, Xu Y, Li B, Wang DW. Applications of the method of high resolution melting analysis for diagnosis of Leber's disease and the three primary mutation spectrum of LHON in the Han Chinese population. Gene. 2013 Jan 1;512(1):108-12. doi: 10.1016/j.gene.2012.09.110. Epub 2012 Oct 9. PMID 23063736
- [Background] Shi H, Gao J, Pei H, Liu R, Hu WK, Wan X, Li T, Li B. Adeno-associated virus-mediated gene delivery of the human ND4 complex I subunit in rabbit eyes. Clin Exp Ophthalmol. 2012 Dec;40(9):888-94. doi: 10.1111/j.1442-9071.2012.02815.x. Epub 2012 Jul 2. PMID 22612072
- [Background] Feuer WJ, Schiffman JC, Davis JL, Porciatti V, Gonzalez P, Koilkonda RD, Yuan H, Lalwani A, Lam BL, Guy J. Gene Therapy for Leber Hereditary Optic Neuropathy: Initial Results. Ophthalmology. 2016 Mar;123(3):558-70. doi: 10.1016/j.ophtha.2015.10.025. Epub 2015 Nov 19. PMID 26606867
- [Background] Erickson RP. Leber's optic atrophy, a possible example of maternal inheritance. Am J Hum Genet. 1972 May;24(3):348-9. No abstract available. PMID 5063796
- [Background] Wallace DC, Singh G, Lott MT, Hodge JA, Schurr TG, Lezza AM, Elsas LJ 2nd, Nikoskelainen EK. Mitochondrial DNA mutation associated with Leber's hereditary optic neuropathy. Science. 1988 Dec 9;242(4884):1427-30. doi: 10.1126/science.3201231.
- [Background] Huoponen K, Vilkki J, Aula P, Nikoskelainen EK, Savontaus ML. A new mtDNA mutation associated with Leber hereditary optic neuroretinopathy. Am J Hum Genet. 1991 Jun;48(6):1147-53. PMID 1674640
- [Background] Mackey D, Howell N. A variant of Leber hereditary optic neuropathy characterized by recovery of vision and by an unusual mitochondrial genetic etiology. Am J Hum Genet. 1992 Dec;51(6):1218-28. PMID 1463007
- [Background] Maguire AM, Simonelli F, Pierce EA, Pugh EN Jr, Mingozzi F, Bennicelli J, Banfi S, Marshall KA, Testa F, Surace EM, Rossi S, Lyubarsky A, Arruda VR, Konkle B, Stone E, Sun J, Jacobs J, Dell'Osso L, Hertle R, Ma JX, Redmond TM, Zhu X, Hauck B, Zelenaia O, Shindler KS, Maguire MG, Wright JF, Volpe NJ, McDonnell JW, Auricchio A, High KA, Bennett J. Safety and efficacy of gene transfer for Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2240-8. doi: 10.1056/NEJMoa0802315. Epub 2008 Apr 27. PMID 18441370
- [Background] Bainbridge JW, Smith AJ, Barker SS, Robbie S, Henderson R, Balaggan K, Viswanathan A, Holder GE, Stockman A, Tyler N, Petersen-Jones S, Bhattacharya SS, Thrasher AJ, Fitzke FW, Carter BJ, Rubin GS, Moore AT, Ali RR. Effect of gene therapy on visual function in Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2231-9. doi: 10.1056/NEJMoa0802268. Epub 2008 Apr 27. PMID 18441371
- [Background] Hauswirth WW, Aleman TS, Kaushal S, Cideciyan AV, Schwartz SB, Wang L, Conlon TJ, Boye SL, Flotte TR, Byrne BJ, Jacobson SG. Treatment of leber congenital amaurosis due to RPE65 mutations by ocular subretinal injection of adeno-associated virus gene vector: short-term results of a phase I trial. Hum Gene Ther. 2008 Oct;19(10):979-90. doi: 10.1089/hum.2008.107. PMID 18774912
- [Background] Hufnagel RB, Ahmed ZM, Correa ZM, Sisk RA. Gene therapy for Leber congenital amaurosis: advances and future directions. Graefes Arch Clin Exp Ophthalmol. 2012 Aug;250(8):1117-28. doi: 10.1007/s00417-012-2028-2. Epub 2012 May 29. PMID 22644094
- [Background] Howell N, Bindoff LA, McCullough DA, Kubacka I, Poulton J, Mackey D, Taylor L, Turnbull DM. Leber hereditary optic neuropathy: identification of the same mitochondrial ND1 mutation in six pedigrees. Am J Hum Genet. 1991 Nov;49(5):939-50. PMID 1928099
- [Background] Zhang Y, Tian Z, Yuan J, Liu C, Liu HL, Ma SQ, Li B. The Progress of Gene Therapy for Leber's Optic Hereditary Neuropathy. Curr Gene Ther. 2017;17(4):320-326. doi: 10.2174/1566523218666171129204926. PMID 29189152
- [Derived] Liu HL, Yuan JJ, Tian Z, Li X, Song L, Li B. What are the characteristics and progression of visual field defects in patients with Leber hereditary optic neuropathy: a prospective single-centre study in China. BMJ Open. 2019 Mar 15;9(3):e025307. doi: 10.1136/bmjopen-2018-025307. PMID 30878986